CLINICAL TRIAL: NCT05224869
Title: A Non-Randomized Phase II Study of the Reduction in Rectal V100 With the Use of Rectal Spacer Hydrogel in the Management of Intermediate Risk Prostate Cancer Treated With Combined Modality Radiation Therapy
Brief Title: Rectal Spacer Hydrogel Before Radiation Therapy in Reducing Radiation Dose to the Rectum in Patients With Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Was not meeting target enrollment; other treatment options precluded completing study
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Richard Stock, Professor, Radiation Oncology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 21-0603
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Brachytherapy; Radioactive Seed implant; Rectal Spacer; SpaceOAR
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Physical Examination; Radiosurgery; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients with prostate cancer (Experimental): Patients undergo hydrogel rectal spacer placement on day 1. Within 2 weeks (+/-1 week) after Rectal Spacer placement, patients will be scheduled for CT simulation for external beam treatment planning. Patients will begin the SBRT of 24Gy in 5 fractions within 2 weeks (+/-1 week) from the simulation date. Within 4 weeks (+/-1 week) of last day of SBRT, patients undergo brachytherapy. Patient will return for post-implant CT-based dosimetry analysis 4 weeks (+/- 1 week) post brachytherapy,
  Interventions: Device: Medical Device Usage and Evaluation; Procedure: CT simulation; Procedure: Stereotactic body radiation therapy; Radiation: Brachytherapy; Procedure: Post-implant dosimetry scan

INTERVENTIONS:
Device: Medical Device Usage and Evaluation — Undergo hydrogel rectal spacer placement
  Other Names: Hydrogel rectal spacer; SpaceOAR Hydrogel
Procedure: CT simulation — CT simulation of radiation treatment planning 2-7 days after hydrogel placement
Procedure: Stereotactic body radiation therapy — SBRT in 5 fractions over 1 week, 7 days after CT simulation
  Other Names: SBRT
Radiation: Brachytherapy — one month after completing SBRT
Procedure: Post-implant dosimetry scan — one month after brachytherapy

SUMMARY:
This phase II trial studies the effect of rectal spacer hydrogel before radiation therapy in reducing radiation dose to the rectum in patients with prostate cancer. Rectal spacer hydrogen is a soft gel material used to create a space between the rectum and prostate during radiation treatment. The rectal spacer gel is made up of 90% water and 10% polyethylene glycol and is injected as a liquid through a needle inserted between the rectum and prostate. It stays in place for about 3 months and is naturally absorbed into the body and removed through urine in about 6 months. By pushing the prostate further from the rectum with the hydrogel, it may help spare the rectum from receiving radiation during standard of care stereotactic body radiation therapy and brachytherapy treatment.

DETAILED DESCRIPTION:
The purpose of this research study is to observe the effects of using an FDA-approved rectal spacer device known as the SpaceOAR Hydrogel, which is a soft gel material used to create a space between the rectum and prostate during radiation treatment. The rectal spacer gel is made up of 90% water and 10% polyethylene glycol and is injected as a liquid through a needle inserted between the rectum and prostate. It will stay in place for about 3 months and is naturally absorbed into the body and removed through urine in about 6 months. By pushing the prostate further from the rectum with the hydrogel, it will help spare the rectum from receiving radiation during the standard of care stereotactic body radiation treatment participant will be receiving, along with the brachytherapy treatment. The hydrogel rectal spacer has been shown to be very safe and effective at reducing radiation dose to the rectum during external radiation treatments, but has not been well-studied when using a combination of Stereotactic Body Radiation Therapy (SBRT) and brachytherapy. The goal of this research is to determine how effective the SpaceOAR hydrogel rectal spacer is at decreasing radiation side effects that can occur in the rectum, which can include discomfort or bleeding. The researchers also want to see how the use of this device affects the doctor's ability to perform the brachytherapy implant safely and effectively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/biopsy confirmed adenocarcinoma of prostate within 1 year of registration
* Disease confined to the prostate. Prostate volume must be <150cc confirmed by pelvic CT (with or without contrast) or pelvic/prostate MRI (with or without contrast) +/- ultrasound, within 8 months of signing research consent
* Age >18
* Patients deemed medically suitable to undergo rectal spacer placement, external beam radiotherapy and brachytherapy at the discretion of the radiation oncologist, urologist, medical oncologist and/or internist.
* ECOG score of 0-2.
* One or more of the following risk factors for intermediate risk prostate cancer; T2b or T2c clinical stage, GS 7 (either 3+4 or 4+3), PSA 10-20.
* Ability to understand and the willingness to sign a written informed consent.
* PSA result within 6 months of simulation

Exclusion Criteria:

* Patients with disease not confined to the prostate based on imaging, biopsy, or clinical exam
* Patients with a prostate size > 100 cc based on computed tomography (CT), magnetic resonance imaging (MRI), or ultrasound measurements
* Patients who have undergone previous rectal, bowel, bladder, or prostate surgeries in the past
* Patients with previous treatments for their prostate cancer or that are currently receiving any other experimental therapies
* Patients who have undergone prior pelvic radiotherapy
* Patients with high risk prostate cancer that have any of the following risk factors; GS >= 8, PSA > 20, clinical or imaging stage T3a or higher
* Patients receiving antiandrogen therapy (ADT)
* Patients with any prior active or treated genitourinary malignancy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
The proportion of participants that achieve V100rectum < 0.75 cc | At 1 month post-brachytherapy (at about 2 months)
  Volume of the rectum receiving at least 100% of the prescribed dose (V100rectum) < 0.75 cc rate will be estimated as the proportion of patients that achieve V100rectum < 0.75 cc at the post-implant dosimetry computed tomography scan 1 month following brachytherapy along with a corresponding two-sided 90% confidence interval using the methods and software introduced by Koyama and Chen which accounts for the group sequential nature of the design

SECONDARY OUTCOMES:
D90prostate | At the time of post-implant dosimetry (at about 3 months)
  Radiation dose covering 90% of the prostate (D90prostate)
V150prostate | At the time of post-implant dosimetry (at about 3 months)
  Volume of the prostate receiving at least 150% of the prescribed dose (V150prostate)
Number of participants with anatomic distortions | At the time of the brachytherapy implant (at about 2 months)
  Degree of anatomic distortions present while using the brachytherapy template assessed by the physician. Will be summarized as N (%) of patients where varying levels of anatomic distortion was present: No Pubic Arch interference, =< 5 mm interference and > 5mm interference.
Number of participants with radiographic distortion | At the time of the brachytherapy implant (at about 2 months)
  Degree of ultrasound distortion present Assessed by the physician. Will be summarized as N (%) of patients where varying levels of radiographic distortion was present: No Distortion, Mild Distortion, and Severe Distortion.
Change in International Prostate Symptom Score (IPSS) | Baseline and up to 2 years post-treatment
  The IPSS endpoint is based on a questionnaire made up of eight items, seven of which measure symptom severity and one which assesses quality of life. The symptom severity items include: feeling of incomplete emptying, frequency, intermittency, urgency, weak stream, straining and nocturia, each of which is rated from 0 (''not at all'') to 5 (''almost always''). The IPSS total score ranges from 0-35, with a higher score representing greater severity of symptoms, which can be further categorized into mild (0-7), moderate (8-19) and severe (20-35) symptom severity.
Change in Sexual Health Index in Men (SHIM) | Baseline and up to 2 years post-treatment
  The SHIM endpoint is based on a questionnaire made up of five questions each of which is rated from 1 (''very low'') to 5 (''very high''). The SHIM total score (calculated by summing the individual rating for each question) ranges from 5-25, with a lower score representing greater severity of symptoms which can be further categorized into severe erectile dysfunction (ED) (5-7), moderate ED (8-11), mild to moderate ED (12-16), mild ED (17-21) and no ED (22-25).
Change in Expanded Prostate Cancer Index Composite (EPIC) | Baseline and up to 2 years post-treatment
  The EPIC endpoint is based on a questionnaire made up of 50 questions assessing the disease specific aspects of prostate cancer and its therapies and comprises four summary domains (Urinary, Bowel, Sexual and Hormonal). Factor analysis supports dividing the Urinary Domain Summary Score into two distinct Incontinence and Irritative/Obstructive subscales (Subscales scored from 0-100). In addition, each Domain Summary Score has measurable Function Subscale and Bother Subscale components. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stock, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Sharing data is not planned unless specifically requested by another institution.

REFERENCES:
- [Background] Nehlsen AD, Sindhu KK, Moshier E, Sfakianos JP, Stock RG. The impact of a rectal hydrogel spacer on dosimetric and toxicity outcomes among patients undergoing combination therapy with external beam radiotherapy and low-dose-rate brachytherapy. Brachytherapy. 2021 Mar-Apr;20(2):296-301. doi: 10.1016/j.brachy.2020.09.018. Epub 2020 Nov 13. PMID 33199175